CLINICAL TRIAL: NCT00768222
Title: Pilot Evaluation of Cosmetic Outcome and Surgical Site Infection Rates of Coated VICRYL* Plus Antibacterial (Polyglactin 910) Suture Compared to Chinese Silk in Scheduled Breast Cancer Surgery
Brief Title: Coated VICRYL* Plus Suture Compared to Chinese Silk in Scheduled Breast Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200-08-002
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: wound healing
MeSH Terms: conditions — Breast Neoplasms | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chinese Silk Suture (Active Comparator): Natural, non-absorbable silk suture made from entwined thread from silkworm larva, commercially available in China, used in a simple interrupted transdermal suture pattern
  Interventions: Device: silk suture
- VICRYL* Plus Suture (Experimental): Synthetic absorbable surgical suture composed of a copolymer of 90% glycolide and 10% L-lactide and containing triclosan antibacterial, used in a subcuticular closure technique
  Interventions: Device: VICRYL* Plus suture

INTERVENTIONS:
Device: silk suture — skin closure
  Other Names: surgical suture (silk)
  Arms: Chinese Silk Suture
Device: VICRYL* Plus suture — skin closure
  Other Names: Polyglactin 910 (Vicryl); Triclosan (antibacterial)
  Arms: VICRYL* Plus Suture

SUMMARY:
This is a 90-day study to evaluate cosmetic outcome and Surgical Site Infection in approximately 100 patients from 6 centers in China undergoing scheduled modified radical mastectomy for breast cancer.

DETAILED DESCRIPTION:
Patients will be evaluated post-procedure on Days 3, 5, 7, 12, 30 and 90 for cosmetic outcome and surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with written informed consent
* Scheduled for a modified radical mastectomy
* Surgical wound classified Class I/Clean using the CDC SSI Surgical Wound Classification

Exclusion Criteria:

* Unable to give consent and unlikely to comply with study requirements and complete the 90-day follow up visit
* Undergoing surgery for modified radical mastectomy with immediate breast reconstruction, cosmetic breast operations, reduction, expansion, insertion of prothesis, duct ectasia or infective breast disease or implant
* Surgical wounds classified as Class II, III or IV using CDC SSI Surgical Wound Classification
* Has inflammatory cancers or skin ulceration
* Has known allergy or intolerance to triclosan
* Has compromised wound healing or chronic immune deficiency, for example diabetes, prolonged steroid use, AIDS or substance abuse
* Has serious heart and/or lung disease
* Has skin scar history or family history
* Has direct relationship to or involvement in this or other studies under the direction of the investigator or center
* Received an experimental drug or device within 30 days prior to the planned start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao ZHANG, MD, Principal Investigator — Capital Medical University Affiliated Beijing Friendship Hospital
Locations (6):
- China (6):
  - Capital Medical Univ. affiliated Hospital, Beijing
  - Jilin Univ. affiliated Second Hospital, Changchun
  - Dalian Medical Univ. affiliated first Hospital, Dalian
  - First Affiliated Hospital, Sun Yat-sen Univ., Guangzhou
  - Fudan Univ. affiliated Zhongshan Hospital, Shanghai
  - Shanghai Jiao Tong Univ. affiliated Ruijin Hospital, Shanghai

REFERENCES:
- [Derived] Zhang ZT, Zhang HW, Fang XD, Wang LM, Li XX, Li YF, Sun XW, Carver J, Simpkins D, Shen J, Weisberg M. Cosmetic outcome and surgical site infection rates of antibacterial absorbable (Polyglactin 910) suture compared to Chinese silk suture in breast cancer surgery: a randomized pilot research. Chin Med J (Engl). 2011 Mar;124(5):719-24. PMID 21518565

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Started | 50 | 51
Completed | 46 | 47
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture | Total
Number analyzed (Participants) | 50 | 51 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.3) | 53.0 (12.1) | 52.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Score on Cosmetic Outcome Visual Analog Scale (VAS)
Description: Post-operative cosmetic outcome assessed on surgical site photographs by an independent blinded central assessor using a validated 100 mm visual analog scale, with 0 representing the worst possible scar and 100 representing the best possible scar
Time Frame: 30 days (+/- 5) post-operative
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 45.4 (12.0) | 67.2 (18.2)

2. Secondary Outcome: Mean Cosmetic Outcome Score on Modified Hollander Scale
Description: Post-operative cosmetic outcome assessed on surgical site by investigator using the modified Hollander Cosmetic Scale (mHCS) with 0 representing worst and 6 representing best, calculated by adding the individual scores on each of 6 categories (step-off borders, contour irregularities, wound margin separation, edge inversion, excessive inflammation, and overall appearance
Time Frame: 12 days
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 5.2 (1.2) | 5.7 (0.8)

3. Secondary Outcome: Mean Cosmetic Outcome Score on Modified Hollander Scale
Description: as for outcome 2
Time Frame: 30 days
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 5.0 (1.2) | 5.7 (0.5)

4. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: Post-operative assessment of wound by trained observer to identify SSI based on several characteristics that are assigned points that contribute to a total score, with 0-10 representing satisfactory healing (best), 11-20 representing disturbance of healing, 21-30 representing minor wound infection, 31-40 representing moderate wound infection, and over 40 representing severe wound infection (worst)
Time Frame: Day 3
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 1.6 (1.3) | 1.2 (1.3)

5. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: as for outcome 4
Time Frame: Day 5
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 1.5 (1.3) | 1.2 (1.4)

6. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: as for outcome 4
Time Frame: Day 7
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 1.4 (1.3) | 0.9 (1.3)

7. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: as for outcome 4
Time Frame: Day 12
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 4.6 (3.6) | 3.3 (3.8)

8. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: as for outcome 4
Time Frame: Day 30
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 4.6 (3.5) | 3.7 (5.2)

9. Secondary Outcome: Mean Surgical Site Infection Score on Modified ASEPSIS Scale
Description: as for outcome 4
Time Frame: Day 90
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Number analyzed (Participants) | 50 | 51
score on scale | 4.3 (3.3) | 3.2 (3.6)

ADVERSE EVENTS:
Time Frame: Intraoperative through 90 days post-operative
Description: Investigators were required to report all adverse events to the sponsor within 24 hours of becoming aware of the event. Subjects were encouraged to report AEs spontaneously or in response to general, non-directed questioning at each of the visits.
Arm/Group | Chinese Silk Suture | VICRYL* Plus Suture
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/51
Other Adverse Events (participants affected / at risk) | 14/50 | 7/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chinese Silk Suture (N=50) | VICRYL* Plus Suture (N=51)
Deep incisional SSI (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Allergic shock (General disorders) | 1 (1) | 0 (0)
Skin lymphangitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow suppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chinese Silk Suture (N=50) | VICRYL* Plus Suture (N=51)
Incision site infection (Infections and infestations) | 4 (4) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Skin necrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other